CLINICAL TRIAL: NCT05970029
Title: Influence of the Communication Between Nursing Staff and Patients on the Analgesic Response Following Caesarean Section
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Haifa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 0014-23-CMC
Record Dates: First submitted 2023-04-20; First posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-04

CONDITIONS: Acute Pain
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Intervention Model Description: Parallel design - subjects are allocated into one of two study arms
Who Masked: Participant, Outcomes Assessor
Masking Description: At the time of analgesic request the nurse will open an envelop in which the participant assignment will be described. While the nurse (the communicator) is not blinded, the participants are blinded. The pain intensity reports will be recoded by the participants via a secured link, hence the participants are also the outcome assessor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced communication (Experimental): In the enhanced communication study arm the nurse will say to the patient: "I will now give you our first line analgesic medication, liquid Dipyrone. It is a very efficient treatment and based on my experience you will very soon feel significant pain relief".
  Interventions: Behavioral: Communication style
- Normal communication (Other): In the normal communication study arm the communication between the nurse and patients will be as usual in clinical practice - i.e. - no instruction are given to the nurses regarding on how to communicate with patients while administrating the treatment.
  Interventions: Behavioral: Communication style

INTERVENTIONS:
Behavioral: Communication style — The verbal communication between the nurse and the patient at the time of analgesic administration

SUMMARY:
Effective management of postoperative pain is a priority for women undergoing cesarean delivery. Despite availability of modern analgesics, postoperative pain management remains a challenge.

One opportunity to enhance the analgesic effect of the pharmacological treatments given to people suffering from pain (and not just pain) is through increasing the expectations for pain relief following treatment. Although much knowledge has been accumulated about the significant effect of expectations on pain, virtually all evidence are based on experimental studies carried out in laboratory settings, and there is a need to investigate how this knowledge could translated into improved clinical care.

The aim of the current study is to examine whether the communication style between the nursing staff and the patient during analgesic administration will affect the results of pain relief treatment in the mother-newborn ward after cesarean section. As another goal, the study will examine whether relevant patient's characteristics will predict the effectiveness of the treatment.

DETAILED DESCRIPTION:
The study will be carried out in the maternity ward at Carmel Hospital. The study population will include patients who are about to undergo an elective caesarean section under spinal anesthesia. The recruitment will be done pre-surgery. Following consent, participants will receive an explanation about how to assess pain and will fill out the research questionnaires. Communication is the independent variable in this study , which has 2 levels - the increased communication arm and the normal communication arm. Each arm will include 40 patients that will be randomly divided between the arms. The dependent variable is the treatment efficacy, based on the changes in the intensity of the patient's pain one hour after the administration of analgesic. The Self-Consciousness Scale (SCS-R) and the Short suggestibility scale (SSS) will be used to assess relevant personality traits.

ELIGIBILITY:
Inclusion Criteria:

* Be able to provide signed and dated written informed consent and to be compliant with the schedule of protocol assessments.
* Females aged 18 till 50
* Undergoing cesarean section

Exclusion Criteria:

* Mental retardation and cognitive impairment

study.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Only woman undergoing cesarian section
Enrollment: 80 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Change in pain intensity on the 0-10 pain scale | one hour
  Change in pain intensity one hour following administration of analgesics

OTHER OUTCOMES:
The Self-Consciousness Scale (SCS-R) | Once, at baseline
  Assessment of direction of attention. Three variables are calculated (private and public attention and social anxiety)
The Short suggestibility scale (SSS) | Once, at baseline
  Assessment of suggestibility score, ranging from 21 to 84, higher scores represent more tendency to suggestibility

CONTACTS AND LOCATIONS:
Overall Officials: Vered Cohen, BA, Principal Investigator — Carmel Medical Center
Locations (1):
- Carmel Medical Center, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No
A link to the data location will be published in the article summarizing the results